CLINICAL TRIAL: NCT07093411
Title: A Phase I, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LUCAR-E9D,LUCAR-E9K, a Dual-targeted Cell Product Targeting CD19/CD20, in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Targeting CD19/CD20 Dual-targeted Cell in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2406-0001
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-06

CONDITIONS: B-cell Non-Hodgkin Lymphoma Recurrent B-cell Non-Hodgkin Lymphoma Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LUCAR-E9D or LUCAR-E9K (Experimental): Each subject will be given a single-dose LUCAR-E9D or LUCAR-E9K cells infusion at each dose level.
  Interventions: Biological: LUCAR-E9D or LUCAR-E9K cells product

INTERVENTIONS:
Biological: LUCAR-E9D or LUCAR-E9K cells product — Prior to infusion of the LUCAR-E9D or LUCAR-E9K cells product subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine

SUMMARY:
A phase I, open-label clinical study to evaluate the safety, tolerability, and efficacy of LUCAR-E9D,LUCAR-E9K, a dual-targeted cell preparation targeting CD19/CD20, in patients with relapsed/refractory B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation/dose extension study to assess the safety, tolerability, and efficacy of LUCAR-E9D,LUCAR-E9K in the patient ≥ 18 years of age with relapsed or refractory B-cell non-Hodgkin lymphoma. Subjects who meet the eligibility criteria will receive a single dose of LUCAR-E9D,LUCAR-E9K injection. The study will include the following sequential phases: screening, pre-treatment (lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures and have signed informed consent.
2. Aged 18-75 years (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed B-cell non-Hodgkin Lymphoma that expresses at least one of CD19/CD20.
5. At least one evaluable tumor lesion according to Lugano 2014 criteria.
6. Response to prior therapy is consistent with one of the following:

1） Patients with B-NHL who are primary refractory and are unsuitable or unwilling to receive autologous CAR-T cell therapy; 2） primary refractory is defined as the best response to first-line treatment being SD or PD; 3） Relapse within 12 months after achieving CR with first-line chemotherapy and immunotherapy; 7. Life expectancy≥ 3 months 8. Women of childbearing potential must have a negative highly sensitive serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening and before the first administration of cyclophosphamide and fludarabine treatment;

Exclusion Criteria:

1. Diagnosed with or treated for other invasive malignancies besides B-cell non-Hodgkin lymphoma.
2. Active acute or chronic graft-versus-host disease (GVHD), except for grade 1 skin involvement; or requiring immunosuppressive treatment for GVHD within 4 weeks prior to enrollment;
3. Active CNS involvement (symptomatic or positive cerebrospinal fluid or imaging data), prior CNS infiltration but currently in remission (asymptomatic and negative cerebrospinal fluid and/or imaging data) is eligible;
4. Significant bleeding tendency, such as gastrointestinal bleeding, hemorrhagic cystitis, coagulopathy.
5. Chronic diseases treated with steroids or other immunosuppressants. The following situations are excluded: use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylaxis;
6. Severe underlying diseases, such as: - Evidence of severe active viral, bacterial infections, or uncontrolled systemic fungal infections; - Active or unstable autoimmune diseases, or autoimmune diseases within the past 3 years with potential for relapse;
7. Breastfeeding women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs (Treatment-emergent Adverse Events) | 2 years after LUCAR-E9D,LUCAR-E9K infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | 2 years after LUCAR-E9D,LUCAR-E9K infusion
  CAR positive T cells and CAR transgene levels in peripheral blood after LUCAR-E9D,LUCAR-E9K infusion.
Pharmacokinetics in bone marrow | 2 years after LUCAR-E9D,LUCAR-E9K infusion
  CAR positive T cells and CAR transgene levels in bone marrow after LUCAR-E9D,LUCAR-E9K infusion.
The recommended Phase II dose (RP2D) for this cell therapy | 30 days after LUCAR-E9D,LUCAR-E9K infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, 2 years after LUCAR-E9D,LUCAR-E9K infusion
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LUCAR-E9D,LUCAR-E9Kcell infusion
Progression-free survival (PFS) | Through study completion, 2 years after LUCAR-E9D,LUCAR-E9K infusion
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LUCAR-E9D, LUCAR-E9K to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Through study completion, 2 years after LUCAR-E9D,LUCAR-E9K infusion
  Overall Survival (OS) is defined as the time from the date of first infusion of LUCAR-E9D,LUCAR-E9Kto death of the subject
Time to Response (TTR) | Through study completion, minimum 2 years after LUCAR-E9D,LUCAR-E9K infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LUCAR-E9D,LUCAR-E9Kto the date of the first response evaluation of the subject who has met all criteria for CR or PR.
Time to Response (TTR) | Through study completion, 2 years after LUCAR-E9D,LUCAR-E9K infusion
  Time to Response (TTR) is defined as the time from the date of first infusion of LUCAR-E9D,LUCAR-E9Kto the date of the first response evaluation of the subject who has met all criteria for CR or PR.
Duration of Response (DoR) | Through study completion, minimum 2 years after LUCAR-E9D,LUCAR-E9K infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or PR) to the first documented relapse evidence of the responders.
Immunogenicity assessment of LUCAR-E9D or LUCAR-E9Kcells | Through study completion, 2 years after LUCAR-E9D,LUCAR-E9K infusion
  The incidence of Anti- LUCAR-E9D or LUCAR-E9Kantibody in patients who received LUCAR-E9D,LUCAR-E9Kcells infusion

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: No